CLINICAL TRIAL: NCT06475209
Title: Observational Study on the Efficacy and Safety of Adebrelimab Combined With Apatinib in Maintenance Therapy for Extensive-Stage Small Cell Lung Cancer
Brief Title: Adebrelimab + Apatinib in SCLC Maintenance Therapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tang-Du Hospital (Other)
Collaborators: Jiangsu Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202404-25
Record Dates: First submitted 2024-06-20; First posted 2024-06-26 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: SCLC
Keywords: SCLC; Adebrelimab; Apatinib; Maintenance Therapy
MeSH Terms: interventions — apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adebrelimab combined with Apatinib (Experimental): Evaluation of the Efficacy and Safety of Adebrelimab in Combination with Apatinib in Maintenance Therapy for Extensive-Stage Small Cell Lung Cancer Each treatment cycle spans 3 weeks. Sequential medication administration begins on the first day of each cycle: Adebrelimab is administered at a dosage of 1200mg on day 1, every 3 weeks, while Apatinib is given orally at a dosage of 250mg daily from day 1 to day 14, every 3 weeks, with a one-week hiatus following two weeks of continuous intake. Administration timing allows for a window of ±5 days. Subjects are required to undergo comprehensive assessments, including vital signs monitoring, anthropometric measurements, physical examinations, laboratory analyses, and performance status evaluations, to assess treatment tolerability for continuation.
  Interventions: Drug: Adebrelimab combined with Apatinib

INTERVENTIONS:
Drug: Adebrelimab combined with Apatinib — Each treatment cycle spans 3 weeks. Sequential medication administration begins on the first day of each cycle: Atezolizumab is administered at a dosage of 1200mg on day 1, every 3 weeks, while Apatinib is given orally at a dosage of 250mg daily from day 1 to day 14, every 3 weeks, with a one-week hiatus following two weeks of continuous intake. Administration timing allows for a window of ±5 days. Subjects are required to undergo comprehensive assessments, including vital signs monitoring, anthropometric measurements, physical examinations, laboratory analyses, and performance status evaluations, to assess treatment tolerability for continuation.

SUMMARY:
This prospective clinical study aims to evaluate and observe the efficacy and safety of Atezolizumab combined with Apatinib in maintenance therapy for extensive-stage small cell lung cancer using a single-arm trial design.

The study is planned to be conducted in Shaanxi Province, China, with an initial target enrollment of 60 patients. The study commenced in February 2024, and recruitment is expected to conclude around December 2025, with the trial anticipated to end by December 2026. Assuming no occurrences such as withdrawal of informed consent by subjects, intolerable adverse drug reactions, or investigator-assessed unsuitability for further participation, each participant's estimated duration of study treatment will continue until radiographically confirmed tumor progression.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary participation with signed informed consent and good compliance for follow-up.
2. Age between 18 and 75 years old.
3. Histologically or cytologically confirmed extensive-stage small cell lung cancer (LS-SCLC) according to the AJCC 8th edition or VALG phase II staging criteria.
4. ECOG performance status score: 0 to 2.
5. Absence of disease progression after receiving 4-6 cycles of platinum-based chemotherapy combined with Atezolizumab induction therapy.
6. Recovery of non-hematologic adverse reactions to grade 1 (except for alopecia, skin pigment changes, or as determined by the investigator) following induction therapy.
7. Time from the end of induction treatment (last dose) to initiation of maintenance treatment ≤ 6 weeks.
8. At least one measurable lesion assessed by the investigator according to RECIST 1.1.
9. Expected life expectancy of at least 3 months.
10. Normal function of major organs, meeting the following criteria:

    * Bone marrow function: Absolute neutrophil count (ANC) ≥ 1.5×10^9/L (grade 1 according to CTCAE 5.0); platelets ≥ 100×10^9/L; hemoglobin > 80g/L.
    * Renal function: Creatinine ≤ 1.5 times the upper limit of normal (ULN), grade 1 according to CTCAE. Note: If creatinine is greater than 1.5 times the ULN, creatinine clearance must be > 50ml/min.
    * Liver function: Bilirubin ≤ 1.5 times ULN (grade 1 according to CTCAE), patients with Gilbert's syndrome bilirubin ≤ 3.0 times ULN; AST and ALT ≤ 3.0×ULN.
    * Coagulation indicators: International normalized ratio (INR) ≤ 1.55 (if the patient is receiving a stable dose of therapeutic warfarin or low molecular weight heparin, INR is usually between 2 and 3), PTT < 1.2 times ULN.
11. Women of childbearing potential must agree to use contraception during the study and for 6 months after the end of the study (such as an intrauterine device, contraceptive pills, or condoms); serum or urine pregnancy test must be negative within 1 week before enrollment, and must be non-lactating patients; men must agree to use contraception during the study and for 6 months after the end of the study.

Exclusion Criteria:

-

Exclusion Criteria:

1. Limited-stage small cell lung cancer (SCLC).
2. Histologically or cytologically confirmed mixed-type SCLC.
3. Prior use of anti-angiogenic drugs or deemed unsuitable for anti-angiogenic therapy by the investigator.
4. Central tumors invading major blood vessels with assessed bleeding risks.
5. Factors affecting oral medication (e.g., dysphagia, chronic diarrhea, intestinal obstruction).
6. Major surgical procedures, incisional biopsies, or significant traumatic injuries within 4 weeks prior to enrollment.
7. Participation in another investigational drug clinical trial within the past 4 weeks.
8. Medical history including:

   * Untreated or symptomatic brain metastases or spinal cord compression.
   * Concurrent active malignant tumors requiring treatment.
   * History of immunodeficiency, including HIV positivity, other acquired or congenital immunodeficiency diseases, or organ transplant recipients.
   * History of substance abuse disorders not amenable to treatment or psychiatric disorders.
9. Presence of any severe and/or uncontrolled diseases including:

   * Poorly controlled hypertension (systolic blood pressure ≥ 150 mmHg, diastolic blood pressure ≥ 100 mmHg).
   * Ischemic heart disease or myocardial infarction of grade I or higher, arrhythmias (including QTc ≥ 450ms for males, QTc ≥ 470ms for females), and ≥ grade 2 congestive heart failure (New York Heart Association [NYHA] functional classification); or left ventricular ejection fraction (LVEF) < 50% based on echocardiography.
   * Decompensated diabetes or other contraindications to high-dose corticosteroid therapy.
   * Worsening chronic obstructive pulmonary disease (COPD) or other severe respiratory diseases requiring hospitalization.
   * Active or uncontrolled severe infections (≥ CTC AE grade 2).
   * Uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage.
   * Liver cirrhosis, decompensated liver disease, active hepatitis, or chronic hepatitis requiring antiviral therapy.
   * Renal insufficiency: Urine protein ≥ ++ on urinalysis, and confirmed 24-hour urine protein quantitation > 1.0 g.
10. Clinically significant hemoptysis (>1/2 teaspoon of fresh blood) or significant bleeding symptoms within the past 3 months prior to enrollment, or evidence of bleeding tendency such as gastrointestinal bleeding, bleeding gastric ulcers, baseline fecal occult blood test ≥ ++, or non-healed wounds, ulcers, or fractures.
11. Occurrence of venous or arterial thrombotic events within the past 6 months prior to enrollment, such as cerebrovascular accidents (including transient ischemic attacks, cerebral hemorrhages, cerebral infarctions), deep vein thrombosis, and pulmonary embolism.
12. Abnormal coagulation function (INR > 1.5 or prothrombin time PT > ULN + 4 seconds or APTT > 1.5 ULN), bleeding tendency, or undergoing thrombolysis or anticoagulant therapy. Use of low-dose heparin (adult daily dose of 0.6-1.2 x 104U) or low-dose aspirin (daily dose ≤ 100 mg) is permitted for prophylactic purposes with INR ≤ 1.5.
13. Patients unable to comply with study procedures, restrictions, and requirements as judged by the investigator are ineligible for participation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-06-20 (Estimated); Primary Completion 2025-12-20 (Estimated); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | Progression-free survival (PFS) analysis based on investigator assessment per RECIST 1.1, and will be assessed up to 2 years
  Progression free survival (PFS) refers to the time from recording the first chemotherapy treatment to the date of disease progression, as assessed by researchers.

SECONDARY OUTCOMES:
Overall Survival | The maximum time from receiving treatment to dying for any reason is 4 years.
  Overall survival (OS) refers to the time that researchers evaluate from recording the first chemotherapy to death (of any cause).
Objective response rate | Data obtained up until progression, or the last evaluable assessment in the absence of progression, will be assessed up to 1 years
  Per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) using Investigator assessments, is defined as the number (%) of patients with response of Complete Response or Partial Response, will be assessed up to 1 years.
Complete Response rate | up to 1 years
  Per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) using Investigator assessments, is defined as the number (%) of patients with response of Complete Response, will be assessed up to 1 years.
Duration of Response | Duration of Response（DoR）analysis based on investigator assessment per RECIST 1.1, and will be assessed up to 1 years
  Duration of Response（DoR）refers to the time from the first assessment as CR or PR to the first assessment as PD or (due to any reason) death

CONTACTS AND LOCATIONS:
Locations (1):
- Tangdu Hospital Affiliated to the Fourth Military Medical University, Xi'an, Shannxi, China